CLINICAL TRIAL: NCT01200381
Title: INvestigation on Routine Follow-up in CONgestive HearT FAilure Patients With Remotely Monitored ICD SysTems
Brief Title: INvestigation on Routine Follow-up in CONgestive HearT FAilure Patients With Remotely Monitored Implanted Cardioverter Defibrillators (ICD) SysTems
Acronym: InContact
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T94
Record Dates: First submitted 2010-09-10; First posted 2010-09-13 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Heart Failure
Keywords: ICD; CRTD; Remote care; Remote monitoring; Heart failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (Active Comparator): Automatic anonymous ICD/CRTD follow up (quarterly remote follow ups)
  Interventions: Other: Quarterly remote follow ups and remote monitoring
- Group B1 (Active Comparator): Personal ICD/CRTD follow up (phone calls + quarterly remote follow ups)
  Interventions: Other: Quarterly remote follow ups + additional phone calls and remote monitoring
- Group B2 (Active Comparator): Personal ICD/CRTD follow up (Quarterly visits)
  Interventions: Other: Quarterly in clinic follow ups and remote monitoring

INTERVENTIONS:
Other: Quarterly remote follow ups and remote monitoring — Quarterly remote follow ups and remote monitoring
  Arms: Group A
Other: Quarterly remote follow ups + additional phone calls and remote monitoring — Quarterly remote follow ups + additional phone calls and remote monitoring
  Arms: Group B1
Other: Quarterly in clinic follow ups and remote monitoring — Quarterly in clinic follow ups and remote monitoring
  Arms: Group B2

SUMMARY:
It's the aim of this study to analyze the benefit of personal patient / physician contacts in heart failure patients with remotely monitored implanted cardioverter defibrillators (ICD) or ICD with cardiac resynchronization therapy (CRT-D).

The personal follow up (in clinic or phone calls) will be compared to completely automatic remote follow ups.

All patients will receive remote monitoring for automatic daily alarm checks and will undergo in clinic follow ups in 12 months intervals

ELIGIBILITY:
Inclusion Criteria:

* Indication for implantation (new, boxchange, upgrade) of ICD/ CRT-D
* Written informed consent
* Ejection Fraction <= 35%
* New York Heart Association (NYHA) Class I-III
* Age >=18 and <=80 years
* In patient's home environment sufficient infrastructure (analog phone line or sufficient strength of GSM (Global System for Mobile communication) mobile phone network) for running a Merlin@home transmitter is available

Exclusion Criteria:

* Arterio ventricular (AV) Block III / AV Block II Type Mobitz
* Severe renal insufficiency
* Coronary angiology intervention within previous 3 months
* Myocardial infarction within previous month
* Life expectancy < 1 year
* Expected poor data quality / compliance
* Pregnancy
* Patient is already participating to another study with active therapy arm

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2010-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Amount of patients with worsened outcome in reference to Packer's "Heart Failure Clinical Composite Response" | 12 months (between 1 and 13 months post implant)

SECONDARY OUTCOMES:
Mortality | 12 months (between 1 and 13 months post implant)
Heart failure hospitalizations | 12 months (between 1 and 13 months post implant)
Cardiovascular events | 12 months (between 1 and 13 months post implant)
Number of additional, unscheduled follow ups | 12 months (between 1 and 13 months post implant)
Number of follow ups with relevant findings | 12 months (between 1 and 13 months post implant)
Number of delivered / appropriate ICD therapies | 12 months (between 1 and 13 months post implant)
Quality of life (MLHFQ) | 12 months (between 1 and 13 months post implant)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Weiss, Prof. Dr. med., Study Chair — Städtisches Klinikum Lüneburg gGmbH
Locations (17):
- Germany (17):
  - SLK-Kliniken Heilbronn GmbH Klinikum am Plattenwald, Bad Friedrichshall
  - Asklepios Klinik Bad Oldesloe, Bad Oldesloe
  - Segeberger Kliniken GmbH, Bad Segeberg
  - Evangelisches Krankenhaus Bielefeld gGmbH, Bielefeld
  - Evangelisches Krankenhaus Kalk, Cologne
  - Universitätsklinikum Essen (AöR), Essen
  - Herzkatheterlabor der Kardiologischen Praxis am Krankenhaus Neu-Bethlehem gGmbH, Göttingen
  - Asklepios Klinik St. Georg, Hamburg
  - Asklepios Klinik Barmbek, Hamburg
  - Klinikum Ingolstadt GmbH, Ingolstadt
  - Kardiologische Praxis - Partnergesellschaft, Ludwigsburg
  - Städtisches Klinikum Lüneburg gGmbH, Lüneburg
  - Marienhaus Klinikum St. Elisabeth-Krankenhaus, Neuwied
  - Praxis Dr. med. Balbach / Ruppert, Nürtingen
  - Kardiologische Gemeinschaftspraxis am Park Sanssouci, Potsdam
  - Klinikum Sindelfingen-Böblingen gGmbH, Sindelfingen
  - Marienhospital Stuttgart, Stuttgart

REFERENCES:
- [Derived] Hansen C, Loges C, Seidl K, Eberhardt F, Troster H, Petrov K, Gronefeld G, Bramlage P, Birkenhauer F, Weiss C. INvestigation on Routine Follow-up in CONgestive HearT FAilure Patients with Remotely Monitored Implanted Cardioverter Defibrillators SysTems (InContact). BMC Cardiovasc Disord. 2018 Jun 28;18(1):131. doi: 10.1186/s12872-018-0864-7. PMID 29954340